CLINICAL TRIAL: NCT04655482
Title: Treat-and-extend Using Aflibercept for Type 3 Neovascularization
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kim's Eye Hospital (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-06-003
Record Dates: First submitted 2020-11-23; First posted 2020-12-07 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Retinal Angiomatous Proliferation
Keywords: Retinal Angiomatous Proliferation; Type 3 neovascularization; Aflibercept; Treat and extend
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Intervention Model Description: Patients diagnosed with type 3 neovascularization Patients treated with treat-and-extend regimen using aflibercept
Masking Description: No masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Patients treated with aflibercept (2.0ml/0.05cc) using treat-and-extend regimen.
  Three monthly loading injections followed by proactive treatment using treat-and-extend regimen. Extension of injection interval by 2 weeks. The maximum injection interval was set as 16 weeks.
  Interventions: Drug: Aflibercept Injection

INTERVENTIONS:
Drug: Aflibercept Injection — Intravitreal injection of aflibercept using treat-and-extend regimen
  :Three monthly loading injections followed by proactive treatment using TAE regimen. Extension of injection interval by 2 weeks. The maximum injection interval was set as 16 weeks.
  Other Names: Intravitreal injection of aflibercept (Eylea, Bayer co.)

SUMMARY:
Type 3 neovascularization is a subtype of neovascular age-related macular degeneration (AMD) that is characterized by intraretinal neovascularization. Treat-and-extend (TAE) regimen is a widely-used, effective anti-vascular endothelial growth factor treatment regimen for neovascular AMD, regardless of subtypes of AMD. The purpose of the present study is to investigate the 18-month treatment outcome of TAE in type 3 neovascularization.

DETAILED DESCRIPTION:
Type 3 neovascularization also called retinal angiomatous proliferation is a subtype of neovascular age-related macular degeneration (AMD) that is characterized by intraretinal neovascularization.

The incidence of type 3 neovascularization is relatively lower than other subtypes of neovascular AMD, constituting 10 to 20% of entire neovascular AMD. However, it is a very important disorder because it often leads bilateral visual deterioration. The high risk of bilateral involvement is characteristic of type 3 neovascularization. In some cases, the visual prognosis of the initially uninvolved eye with better vision, is poorer than the initially involved eye. In addition, profound visual loss may occur during the treatment course, especially in undertreated cases. Thus, preserving vision is particularly important in type 3 neovascularization, which subsequently highlights the importance of investigating more effective treatment strategies. Previous study suggested the need for proactive treatment in type 3 neovascularization to reduce the risk of abrupt visual loss.

Treat-and-extend (TAE) regimen is a widely-used, effective anti-vascular endothelial growth factor treatment regimen for neovascular age-related macular degeneration (AMD), regardless of subtypes of AMD. However, since type 3 neovascularization is at high risk of GA, there has been some debate regarding the benefit of TAE, when compared to the as-needed regimen, for treating type 3 neovascularization. Despite some controversy, reports indicated that increased injection frequency is associated with development or progression of GA. Thus, it is important to balance efficacy and efficiency when treating type 3 neovascularization.

Type 3 neovascularization is a disorder in which the treatment outcome of TAE regimen was first reported. Nevertheless, only limited evidence has been available regarding the efficacy of TAE using aflibercept in this disorder. In addition, all the previous studies were retrospective, based on relatively small study population. Moreover, results of extending the injection interval to 4 months have not yet been reported. Recently, ALTAIR study provides a scientific evidence that injection interval can be extended to 4 months when using TAE regimen. In type 3 neovascularization, extending the injection interval is not only decreases treatment burden of the patient, but also may improve long-term visual outcomes because it may decrease the injection frequency. If this regimen is found to be effective in type 3 neovascularization, it may contribute to more widespread use of TAE regimen using aflibercept for type 3 neovascularization.

In addition, there are two questions which have not been addressed in previous TAE studies for type 3 neovascularization. The first question is "Is the treatment using TAE regimen can impede the fundamental progression of the disorder?". Since visual loss in type 3 neovascularization usually develops in stage 3 disorder (eyes exhibits serous pigment epithelial detachment on OCT, it will be a very meaningful result if TAE can impede stage progression. The second question is "Is there any clues to predict the recurrence of fluid?" Since avoiding under-treatment is very important in type 3 neovascularization, it is very important to identify any factor predictive of recurrence. To address this question, it is necessary to evaluate the serial changes in vascular morphology of type 3 neovascularization lesion. Previously, however, this kind of approach cannot be performed because it requires frequent, serial indocyanine-green angiography examination. Fortunately, recent advent of OCT-angiography provides simple and safe evaluation of vascular morphology. By using OCT-angiography, any vascular morphologic changes preceding the recurrence of fluid during the TAE treatment can be evaluated.

The purpose of the present study is to investigate the 18-month treatment outcome of TAE in type 3 neovascularization. The maximum injection interval was set as 4 months. Since the ALTAIR study nicely show how to extend the interval to 4 months, the study protocol of ALTAIR study was partly adopted in the present study.

ELIGIBILITY:
Inclusion Criteria:

* Willing, committed, and able to return for ALL clinic visits and complete all study related procedures.
* Able to read, (or, if unable to read due to visual impairment, be read to verbatim by the person administering the informed consent or a family member) understand and willing to sign the informed consent form.
* Signed informed consent
* Patients aged 50 years or older
* Patients diagnosed with treatment naïve type 3 neovascularization
* ETDRS BCVA letter score ≥25 letters (approximately 20/320 or better) in the study eye

Exclusion Criteria:

* Any prior ocular (in the study eye) or systemic treatment or surgery for neovascular AMD except dietary supplements or vitamins.
* Prior treatment with anti-VEGF agents
* Known serious allergy to the fluorescein sodium for injection in angiography.
* Significant media opacities, including cataract, in the study eye that might interfere with visual acuity, assessment of safety, or fundus photography.
* Any concurrent ocular condition in the study eye which, in the opinion of the investigator, could either increase the risk to the patient beyond what is to be expected from standard procedures of intraocular injection, or which otherwise may interfere with the injection procedure or with evaluation of efficacy or safety.
* Any ocular or periocular infection within the last 2 weeks prior to Screening in either eye.
* Any history of uveitis in either eye.
* Presence of definite chorioretional anastomosis
* Subretinal hemorrhage that is either 50% or more of the total lesion area, or if the blood is under the fovea and is 1 or more disc areas in size in the study eye. (If the blood is under the fovea, then the fovea must be surrounded 270 degrees by visible CNV.)
* Scar or fibrosis, making up > 50% of total lesion in the study eye.
* Scar, fibrosis, or atrophy involving the center of the fovea in the study eye.
* Presence of retinal pigment epithelial tears or rips involving the macula in the study eye.
* History or clinical evidence of diabetic retinopathy, diabetic macular edema or any other vascular disease affecting the retina, other than AMD, in either eye.
* Any concurrent intraocular condition in the study eye (e.g. cataract) that, in the opinion of the investigator, could require either medical or surgical intervention during the 76 week study period.
* Prior vitrectomy in the study eye
* Any history of macular hole of stage 2 and above in the study eye.
* Any intraocular or periocular surgery within 3 months of Day 1 on the study eye, except lid surgery, which may not have taken place within 1 month of day 1, as long as its unlikely to interfere with the injection.
* Prior trabeculectomy or other filtration surgery in the study eye.
* Uncontrolled glaucoma (defined as intraocular pressure ≥ 25 mmHg despite treatment with antiglaucoma medication) in the study eye.
* Active intraocular inflammation in either eye.
* Active ocular or periocular infection in either eye.
* Aphakia or pseudophakia with absence of posterior capsule (unless it occurred as a result of a yttrium aluminum garnet [YAG] posterior capsulotomy) in the study eye.
* History of corneal transplant or corneal dystrophy in the study eye.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-12-20 (Estimated); Study Completion 2024-08-20 (Estimated)

PRIMARY OUTCOMES:
Change in best-corrected visual acuity (BCVA) | From baseline to week 76
  Change in early treatment of diabetic retinopathy score (ETDRS) BCVA from baseline to week 76

SECONDARY OUTCOMES:
Proportion of patients who gain ≥15 ETDRS letters | from baseline to week 52 and 76
  Measuring proportion of patients who gain ≥15 ETDRS letters
Proportion of patients who loss ≥15 ETDRS letters | from baseline to week 52 and 76
  Measuring proportion of patients who loss ≥15 ETDRS letters
Change in BCVA to wee 52 (interim analysis) | from baseline to week 52
  Change in ETDRS BCVA
Change in central retinal thickness | from baseline to week 52 and 76
  Change in central retinal thickness measured using optical coherence tomography
Proportion of patients without fluid or hemorrhage | at week 52 and 76
  The presence of fluid or hemorrhage is estimated using fundus photographs and optical coherence tomography images
Incidence of geographic atrophy | at baseline, and at weeks 52 and 76
  Geographic atrophy is idenfitied using fundus photographs and optical coherence tomography images
Changes in size of geographic atrophy | from baseline to week 52 and 76
  Changes in size of geographic atrophy is estimated using fundus photographs and optical coherence tomography images
Number of injections | up to week 52 and 76
  Number of injections were counted
The maximum treatment interval and the maximum next planned interval | during week 52 and 76
  The maximum treatment interval and the maximum next planned interval of assessment at the last injection
Proportion of patients showing fovea-involving geographic atrophy or fibrotic scar | at week 52 and 76
  Fovea-involving geographic atrophy or fibrotic scar are idenfitied using fundus photographs and optical coherence tomography images
Proportion of patients showing progression of stages of type 3 neovascularization | Through study completion, 72 weeks
  Progress of disese stages are estimated using optical coherence tomography angiography images
Proportion of patients showing tear of retinal pigment epithelium or subretinal hemorrhage | Through study completion, 72 weeks
  Tear of retinal pigment epithelium or subretinal hemorrhage are idenfitied using fundus photographs and optical coherence tomography images
Morphologic features of type 3 lesion | Through study completion, 72 weeks
  Morphologic features of type 3 lesions are estimated using optical coherence tomography angiography images

CONTACTS AND LOCATIONS:
Overall Officials: Jae Hui Kim, M.D., Principal Investigator — Kim's Eye Hospital, Seoul, South Korea
Locations (1):
- Jae Hui Kim, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Freund KB, Ho IV, Barbazetto IA, Koizumi H, Laud K, Ferrara D, Matsumoto Y, Sorenson JA, Yannuzzi L. Type 3 neovascularization: the expanded spectrum of retinal angiomatous proliferation. Retina. 2008 Feb;28(2):201-11. doi: 10.1097/IAE.0b013e3181669504. PMID 18301024
- [Result] Yannuzzi LA, Negrao S, Iida T, Carvalho C, Rodriguez-Coleman H, Slakter J, Freund KB, Sorenson J, Orlock D, Borodoker N. Retinal angiomatous proliferation in age-related macular degeneration. Retina. 2001;21(5):416-34. doi: 10.1097/00006982-200110000-00003. PMID 11642370
- [Result] Gross NE, Aizman A, Brucker A, Klancnik JM Jr, Yannuzzi LA. Nature and risk of neovascularization in the fellow eye of patients with unilateral retinal angiomatous proliferation. Retina. 2005 Sep;25(6):713-8. doi: 10.1097/00006982-200509000-00005. PMID 16141858
- [Result] Chang YS, Kim JH, Yoo SJ, Lew YJ, Kim J. Fellow-eye neovascularization in unilateral retinal angiomatous proliferation in a Korean population. Acta Ophthalmol. 2016 Feb;94(1):e49-53. doi: 10.1111/aos.12748. Epub 2015 May 17. PMID 25981599
- [Result] Kim JH, Chang YS, Kim JW, Kim CG, Lee DW, Kim HS. LONG-TERM VISUAL CHANGES IN INITIALLY STRONGER FELLOW EYES IN PATIENTS WITH UNILATERAL TYPE 3 NEOVASCULARIZATION. Retina. 2019 Sep;39(9):1672-1681. doi: 10.1097/IAE.0000000000002239. PMID 29979454
- [Result] Kim JH, Chang YS, Kim JW, Kim CG, Lee DW. Early Recurrent Hemorrhage in Submacular Hemorrhage Secondary to Type 3 Neovascularization or Retinal Angiomatous Proliferation: Incidence and Influence on Visual Prognosis. Semin Ophthalmol. 2018;33(6):820-828. doi: 10.1080/08820538.2018.1511814. Epub 2018 Aug 23. PMID 30136868
- [Result] Kim JH, Chang YS, Kim JW, Kim CG, Lee DW. Abrupt visual loss during anti-vascular endothelial growth factor treatment for type 3 neovascularization. Int J Ophthalmol. 2019 Mar 18;12(3):480-487. doi: 10.18240/ijo.2019.03.20. eCollection 2019. PMID 30918819
- [Result] Kim JH, Chang YS, Kim JW, Kim CG, Lee DW. Prechoroidal Cleft in Type 3 Neovascularization: Incidence, Timing, and Its Association with Visual Outcome. J Ophthalmol. 2018 Nov 19;2018:2578349. doi: 10.1155/2018/2578349. eCollection 2018. PMID 30581602
- [Result] Freund KB, Korobelnik JF, Devenyi R, Framme C, Galic J, Herbert E, Hoerauf H, Lanzetta P, Michels S, Mitchell P, Mones J, Regillo C, Tadayoni R, Talks J, Wolf S. TREAT-AND-EXTEND REGIMENS WITH ANTI-VEGF AGENTS IN RETINAL DISEASES: A Literature Review and Consensus Recommendations. Retina. 2015 Aug;35(8):1489-506. doi: 10.1097/IAE.0000000000000627. PMID 26076215
- [Result] Grunwald JE, Daniel E, Huang J, Ying GS, Maguire MG, Toth CA, Jaffe GJ, Fine SL, Blodi B, Klein ML, Martin AA, Hagstrom SA, Martin DF; CATT Research Group. Risk of geographic atrophy in the comparison of age-related macular degeneration treatments trials. Ophthalmology. 2014 Jan;121(1):150-161. doi: 10.1016/j.ophtha.2013.08.015. Epub 2013 Sep 29. PMID 24084496
- [Result] Abdelfattah NS, Al-Sheikh M, Pitetta S, Mousa A, Sadda SR, Wykoff CC; Treat-and-Extend Age-Related Macular Degeneration Study Group. Macular Atrophy in Neovascular Age-Related Macular Degeneration with Monthly versus Treat-and-Extend Ranibizumab: Findings from the TREX-AMD Trial. Ophthalmology. 2017 Feb;124(2):215-223. doi: 10.1016/j.ophtha.2016.10.002. Epub 2016 Nov 15. PMID 27863845
- [Result] Grunwald JE, Pistilli M, Ying GS, Maguire MG, Daniel E, Martin DF; Comparison of Age-related Macular Degeneration Treatments Trials Research Group. Growth of geographic atrophy in the comparison of age-related macular degeneration treatments trials. Ophthalmology. 2015 Apr;122(4):809-16. doi: 10.1016/j.ophtha.2014.11.007. Epub 2014 Dec 24. PMID 25542520
- [Result] Engelbert M, Zweifel SA, Freund KB. "Treat and extend" dosing of intravitreal antivascular endothelial growth factor therapy for type 3 neovascularization/retinal angiomatous proliferation. Retina. 2009 Nov-Dec;29(10):1424-31. doi: 10.1097/IAE.0b013e3181bfbd46. PMID 19898180
- [Result] Castro-Navarro V, Cervera-Taulet E, Montero-Hernandez J, Navarro-Palop C. One-Year Outcomes of the Treat-and-Extend Approach with Aflibercept in Age-Related Macular Degeneration: Effects on Typical Choroidal Neovascularization and Retinal Angiomatous Proliferation. Ophthalmologica. 2016;236(4):215-222. doi: 10.1159/000453281. Epub 2016 Dec 21. PMID 27997921
- [Result] Matsumoto H, Morimoto M, Mimura K, Ito A, Akiyama H. Treat-and-Extend Regimen with Aflibercept for Neovascular Age-Related Macular Degeneration: Efficacy and Macular Atrophy Development. Ophthalmol Retina. 2018 May;2(5):462-468. doi: 10.1016/j.oret.2017.09.002. Epub 2017 Nov 13. PMID 31047326
- [Result] Matsumoto H, Sato T, Morimoto M, Mukai R, Takahashi M, Hiroe T, Ehara K, Takayama M, Mimura K, Kishi S. TREAT-AND-EXTEND REGIMEN WITH AFLIBERCEPT FOR RETINAL ANGIOMATOUS PROLIFERATION. Retina. 2016 Dec;36(12):2282-2289. doi: 10.1097/IAE.0000000000001104. PMID 27336229
- [Result] Su D, Lin S, Phasukkijwatana N, Chen X, Tan A, Freund KB, Sarraf D. AN UPDATED STAGING SYSTEM OF TYPE 3 NEOVASCULARIZATION USING SPECTRAL DOMAIN OPTICAL COHERENCE TOMOGRAPHY. Retina. 2016 Dec;36 Suppl 1:S40-S49. doi: 10.1097/IAE.0000000000001268. PMID 28005662
- [Result] Lee JH, Lee MY, Lee WK. Incidence and risk factors of massive subretinal hemorrhage in retinal angiomatous proliferation. PLoS One. 2017 Oct 12;12(10):e0186272. doi: 10.1371/journal.pone.0186272. eCollection 2017. PMID 29023498
- [Result] Kim JH, Kim JW, Kim CG, Lee DW. Focal retinal pigment epithelium atrophy at the location of type 3 neovascularization lesion: a morphologic feature associated with low reactivation rate and favorable prognosis. Graefes Arch Clin Exp Ophthalmol. 2019 Aug;257(8):1661-1669. doi: 10.1007/s00417-019-04373-4. Epub 2019 May 29. PMID 31144056